CLINICAL TRIAL: NCT04299035
Title: Erector Spinae Plane Block Versus Traditional Pain Management for Enhanced Recovery After Surgery
Brief Title: ESP Block vs. Traditional Pain Management for ERAS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Dmitry Natanel MD, Dr., Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0355-19-SOR
Record Dates: First submitted 2020-03-05; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Erector spinae plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Thoracic surgery + ESPblock (Experimental): Thoracic surgery + ESPblock + standard pain management
  Interventions: Procedure: Erector spinae plane block
- Abdominal surgery + ESPblock (Experimental): Abdominal surgery + ESPblock + standard pain management
  Interventions: Procedure: Erector spinae plane block
- Spinal surgery + ESPblock (Experimental): Spinal surgery + ESPblock + standard pain management
  Interventions: Procedure: Erector spinae plane block
- Thoracic surgery (No Intervention): Thoracic surgery + standard pain management
- Abdominal surgery (No Intervention): Abdominal surgery + standard pain management
- Spinal surgery (No Intervention): Spinal surgery + standard pain management

INTERVENTIONS:
Procedure: Erector spinae plane block — Erector spinae plane block
  Arms: Abdominal surgery + ESPblock; Spinal surgery + ESPblock; Thoracic surgery + ESPblock

SUMMARY:
Patients undergoing thoracotomy, thoracoscopy or other surgical procedures involving the integrity of the chest wall are always in a special point of interest of both surgical and anesthesiological specialities. Most of the patients will describe the pain after thoracic surgery as severe. It might lead to a number of serious complications: respiratory failure due to splinting; inability to clear secretions by effective coughing, with resulting pneumonia; and turning into a chronic pain: the post-thoracotomy pain syndrome.

Traditional pain management in these groups of patients - such as opiate treatment, thoracic epidural analgesia, and non-opioid drugs - may have serious side effects. Large doses of opiates suppress the cough reflex and lead to respiratory depression with subsequent re-intubation and re-ventilation. Thoracic epidural analgesia, though being considered paramount among other analgesic options, requires a significant clinical experience. Still, it might be insufficient for satisfactory pain control and even complicated with pneumothorax, total spinal anaesthesia and inadvertent intravascular injection. Non-steroidal anti-inflammatory drugs (NSAIDs) and Tramadol are weak analgesics inadequate for severe pain control and might be responsible for gastrointestinal bleeding.

We suggest performing erector spinae plane block for intraoperative and postoperative pain management due to the ease of use and better analgesic effect. What remains is hard proof for the clinical efficacy and safety of this block, followed by a demonstration of the uptake of it in the hands of non-regional anaesthetists.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive adult patients who undergo thoracic, spinal or abdominal surgery in Soroka Medical Center, and agree to participate in the study, older than 18 years, who meet criteria of ASA physical status I-II-III-IV class.

Exclusion Criteria:

* Unconscious or mentally incompetent patients or those who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2021-03-05 (Estimated); Study Completion 2021-09-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Pain Score | 3 days
  Reported immediate postoperative VAS score, up to 3rd day
Total pain med consumption in the PACU | 3 hours
  Total Morphine, NSAIDs and Tramadol amount (mg) in the PACU
Length of stay in the PACU | 24 hours
  Length of stay in postoperative care room

SECONDARY OUTCOMES:
Length of hospital stay | 30 days
  Length of hospital stay
Chronic pain development | 6 months
  Rate of chronic pain at 3 and 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dubilet, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- SorokaUMC, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No